CLINICAL TRIAL: NCT02162758
Title: A Randomized, Double-Blind, Phase 4 Study to Evaluate the Effect of Dexlansoprazole 60 mg QD and 60 mg BID on Recurrence of Intestinal Metaplasia in Subjects Who Have Achieved Complete Eradication of Barrett's Esophagus With Radiofrequency Ablation
Brief Title: Effect of Dexlansoprazole 60 mg QD and 60 mg BID on Recurrence of Intestinal Metaplasia in Subjects Who Have Achieved Complete Eradication of Barrett's Esophagus With Radiofrequency Ablation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business Decisions; No Safety Concerns
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DEX-P4-003; U1111-1152-6767 (Registry Identifier: WHO)
Record Dates: First submitted 2014-06-10; First posted 2014-06-13 (Estimated); Results first posted 2017-05-11 (Actual); Last update posted 2017-05-11 (Actual); Status verified 2017-03

CONDITIONS: Barrett's Esophagus
Keywords: Drug therapy
MeSH Terms: conditions — Barrett Esophagus | interventions — Dexlansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexlansoprazole 60 milligram (mg) QD (Experimental): Dexlansoprazole 60 mg, delayed-release capsules, orally, QD and dexlansoprazole 60 mg placebo-matching capsules, orally, once daily for up to 12 months.
  Interventions: Drug: Dexlansoprazole; Drug: Dexlansoprazole Placebo
- Dexlansoprazole 60 mg BID (Experimental): Dexlansoprazole 60 mg, delayed-release capsules, orally, BID for up to 12 months.
  Interventions: Drug: Dexlansoprazole

INTERVENTIONS:
Drug: Dexlansoprazole — Dexlansoprazole delayed-release capsules
  Other Names: Dexilant
Drug: Dexlansoprazole Placebo — Dexlansoprazole placebo-matching capsules
  Arms: Dexlansoprazole 60 milligram (mg) QD

SUMMARY:
This study is designed to evaluate the effect of dexlansoprazole once daily (QD) and twice daily (BID) dosing on the recurrence of intestinal metaplasia (IM) in participants who achieved complete eradication of Barrett's esophagus (BE) with high-grade dysplasia (HGD) following radiofrequency ablation (RFA).

DETAILED DESCRIPTION:
The drug being tested in this study is called dexlansoprazole. The purpose of this study is to evaluate the effect of 12 months of treatment with dexlansoprazole 60 mg QD or dexlansoprazole 60 mg BID on the recurrence of IM in participants who have achieved complete eradication of intestinal metaplasia (CEIM) and dysplasia (CED) with RFA. The study will enroll approximately 150 participants. Participants will be randomly assigned (by chance, like flipping a coin) to one of the two treatment groups which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* Dexlansoprazole 60 mg once a day and placebo (this is a capsule that looks like the study drug but has no active ingredient) once a day
* Dexlansoprazole 60 mg twice a day.

All participants will be asked to take one capsule twice a day at the same time each day throughout the study.

This randomized, double-blind, multi-center, parallel group trial will be conducted in North America. The overall time to participate in this study is up to 13 months. Participants will make 5 visits to the clinic, and will undergo a safety follow-up assessment 30 days after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Is male or female and aged 18 to 80 years, inclusive.
2. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
3. The participant or, when applicable, the participant's legally acceptable representative signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
4. Has a history of initial CEIM following radiofrequency ablation (RFA) for Barrett's esophagus with high-grade dysplasia or low grade dysplasia within the past 3 years.
5. Had attained CEIM within 18 months of receiving his or her first RFA treatment.
6. Has endoscopic and histologic confirmed evidence of CEIM prior to randomization.
7. A male participant who is nonsterilized and sexually active with a female partner of childbearing potential agrees to use adequate contraception from signing of informed consent throughout the duration of the study and for 12 weeks after last dose.
8. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study.

Exclusion Criteria:

1. Has evidence of cardiovascular, pulmonary, central nervous system, hepatic, hematopoietic, renal, metabolic, endocrine or gastrointestinal disease, or serious allergy, asthma, or allergic skin rash that suggests clinically significant, uncontrolled underlying disease or condition (other than the disease being studied), which may impact the ability of the participant to participate or potentially confound the study results.
2. Had previous ablative therapy with a modality other than RFA for Barrett's esophagus (photodynamic therapy, multipolar electrical coagulation, argon plasma coagulation, or laser treatment) with the exception of up to 3 treatments of thermal/coagulation therapy for focal residual disease following otherwise successful RFA therapy.
3. Has a co-existing disease affecting the esophagus (example, erosive esophagitis, esophageal varices, scleroderma, viral or fungal infection, or esophageal stricture), history of radiation therapy or cryotherapy to the esophagus, caustic or physiochemical trauma such as sclerotherapy to the esophagus.
4. Has a known history of eosinophilic esophagitis or endoscopic findings suggestive of eosinophilic esophagitis.
5. Has active gastric or duodenal ulcers within 4 weeks prior to Day -1.
6. Has any finding in his/her medical history, physical examination, or safety clinical laboratory tests giving reasonable suspicion of underlying disease that might interfere with the conduct of the trial.
7. Has a history of hypersensitivity or allergies to dexlansoprazole or any component of dexlansoprazole or any proton pump inhibitor (PPI) (including lansoprazole, omeprazole, rabeprazole, pantoprazole, or esomeprazole) or antacid.
8. Is required to take excluded medications or it is anticipated that the participant will require treatment with at least one of the disallowed concomitant medications during the study evaluation period as specified in the Excluded Medications and Treatments Section..
9. Has a history of malignant disease (except basal cell carcinoma) within 5 years prior to Screening.
10. Has a condition that may require inpatient surgery during the course of the study.
11. Requires dilatation of esophageal strictures and/or strictures preventing passage of the endoscope during the Screening endoscopy. Schatzki's ring (a ring of mucosal tissue near the lower esophageal sphincter) is acceptable.
12. Is known to have acquired immunodeficiency syndrome.
13. Has current or clinical history of Zollinger-Ellison syndrome or other hypersecretory condition.
14. Has a history of gastric, duodenal or esophageal surgery except simple oversew of an ulcer. A history of gastric tube and/or percutaneous endoscopic gastrostomy (PEG) placement is allowed.
15. Had an acute upper gastrointestinal hemorrhage within 4 weeks prior to endoscopy.
16. Has donated or lost greater than or equal to (>=)300 milliliter (mL) blood volume, undergone plasmapheresis, or has had a transfusion of any blood product within 90 days prior to the first dose of study drug.
17. Has a known history of alcohol abuse or illegal drug use within the past 12 months prior to the first dose of study drug, or is unwilling to agree to abstain from alcohol or illegal drug use throughout the study.
18. If female, the participant is pregnant or lactating or intending to become pregnant before, during or within 30 days after last dose of study medication; or intending to donate ova during such time period.
19. If male, the participant intends to donate sperm during the course of this study or within 30 days after last dose of study drug.
20. Is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in the conduct of this study or may consent and assent under duress. Students of the institution/research facility who are under the supervision of, or in a subordinate role to, the investigator are also ineligible.
21. In the opinion of the investigator, is unlikely to comply with the protocol requirements or is unsuitable for any other reason.
22. Has been previously randomized in this study and received at least one dose of double blind study drug treatment.
23. Has received any investigational compound within 30 days prior to Screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-07; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (3):
- United States (3):
  - Jacksonville, Florida
  - Chapel Hill, North Carolina
  - Knoxville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the United States from 16 July 2014 to 09 May 2016.
Pre-assignment Details: Participants with a diagnosis of Barrett's esophagus (BE) who had achieved complete eradication of intestinal metaplasia (CEIM) with radiofrequency ablation (RFA) were enrolled in 1 of the 2 treatment groups: Dexlansoprazole 60 milligram (mg), once-daily (QD); Dexlansoprazole 60 mg, twice daily (BID).
Groups:
- Dexlansoprazole 60 mg QD: Dexlansoprazole 60 mg, delayed-release capsules, orally, QD and dexlansoprazole placebo-matching capsules, orally, QD for up to 12 months.
- Dexlansoprazole 60 mg BID: Dexlansoprazole 60 mg, capsules, orally, BID for up to 12 months.
Period: Overall Study
Arm/Group | Dexlansoprazole 60 mg QD | Dexlansoprazole 60 mg BID
Started | 3 | 3
Completed | 3 | 2
Not Completed | 0 | 1
Not completed — Study termination | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety set included all participants who were randomized and received 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dexlansoprazole 60 mg QD | Dexlansoprazole 60 mg BID | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (8.50) | 67.7 (6.81) | 69.0 (7.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 2 | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic or Latino | 3 | 3 | 6
Race/Ethnicity, Customized [Number; unit: participants]
  White | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 179.3 (4.04) | 167.3 (15.53) | 173.3 (12.09)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 96.80 (20.264) | 88.83 (8.170) | 92.82 (14.491)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 29.95 (4.992) | 31.93 (3.212) | 30.94 (3.908)
Smoking History [Number; unit: participants]
  Never smoked | 1 | 0 | 1
  Ever smoked | 2 | 3 | 5
Number of Smoking Years for Ever Smoked [Number; unit: participants] — Baseline measure was analyzed for those participants who have ever smoked tobacco.
  participants
    16-20 years | 1 | 1 | 2
    Greater than (>) 20 years | 1 | 2 | 3
Current Smoking Status [Number; unit: participants]
  Non smoker | 2 | 3 | 5
  Smoker | 1 | 0 | 1
Number of Packs Per Year [Number; unit: participants] — Baseline measure was analyzed in the participants who currently or have ever smoked tobacco.
  participants
    101-200 packs | 1 | 0 | 1
    301-400 packs | 1 | 0 | 1
    >400 packs | 0 | 1 | 1
    Unknown | 0 | 2 | 2
Alcohol History [Number; unit: participants]
  Never drank alcohol | 2 | 1 | 3
  Drank alcohol | 1 | 2 | 3
Number of Drinking Years [Number; unit: participants] — Baseline measure was analyzed for those participants who currently or have ever drank alcohol.
  participants
    >20 years | 0 | 1 | 1
    Unknown | 1 | 1 | 2
Number of Drinks Per Week [Number; unit: participants] — Baseline measure was analyzed for those participants who currently or have ever drank alcohol.
  participants
    0-5 drinks | 0 | 1 | 1
    6-10 drinks | 0 | 1 | 1
    >30 drinks | 1 | 0 | 1
Current Alcohol Status [Number; unit: participants]
  Current drinker | 0 | 2 | 2
  Non-drinker | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Recurrence of Intestinal Metaplasia (IM)
Description: Recurrence of IM was defined as an esophageal biopsy result indicating BE with or without dysplasia.
Time Frame: Month 12
Population: The Intent-to-treat (ITT) population where Month 12 esophageal biopsy assessment was available. The ITT population included all randomized participants who had documented CEIM at screening and took at least 1 dose of study drug during the treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Dexlansoprazole 60 mg QD | Dexlansoprazole 60 mg BID
Number analyzed (Participants) | 3 | 2
percentage of participants | 0 | 50

2. Secondary Outcome: Percentage of Participants With Recurrence of IM With Dysplasia
Description: Recurrence of IM with dysplasia was defined as an esophageal biopsy result indicating BE with dysplasia.
Time Frame: Month 12
Population: The ITT population where Month 12 esophageal biopsy assessment was available. The ITT population included all randomized participants who had documented CEIM at screening and took at least 1 dose of study drug during the treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Dexlansoprazole 60 mg QD | Dexlansoprazole 60 mg BID
Number analyzed (Participants) | 3 | 2
percentage of participants | 0 | 0

3. Secondary Outcome: Percentage of Participants With Erosive Esophagitis (EE)
Description: The severity of EE was classified into following grades: Grade A: one or more mucosal breaks no longer than 5 millimeter (mm), none of which extends between the tops of the mucosal folds; Grade B: one or more mucosal breaks more than 5 mm long, none of which extends between the tops of two mucosal folds; Grade C: mucosal breaks that extend between the tops of two or more mucosal folds, but which involve less than 75 percent (%) of the esophageal circumference; Grade D: mucosal breaks which involve at least 75% of the esophageal circumference.
Time Frame: Baseline up to Month 12
Population: The ITT population where EE assessment was available. The ITT population included all randomized participants who had documented CEIM at screening and took at least 1 dose of study drug during the treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Dexlansoprazole 60 mg QD | Dexlansoprazole 60 mg BID
Number analyzed (Participants) | 3 | 2
percentage of participants | 0 | 0

4. Secondary Outcome: Change From Baseline in the Gastroesophageal Reflux Disease-Health Related Quality of Life (GERD-HRQL) Total Score
Description: The GERD-HRQL score consisted of 10 questions, where participants were required to answer each question on a scale of 0 to 5 (0: no symptoms; 1: symptoms noticeable but not bothersome; 2: symptoms noticeable and bothersome but not every day; 3: symptoms bothersome every day; 4: symptoms affect daily activity; 5: symptoms are incapacitating to do daily activities). The total score was derived by simply adding the individual score of each question. The total score ranged from 0 to 50 where a higher score indicated more severe disease. The best possible total GERD-HRQL score was 0 (asymptomatic in all questions) and the worst possible score is 50 (incapacitated in all questions).
Time Frame: Baseline and Month 12
Population: The ITT population included all randomized participants who had documented CEIM at screening and took at least 1 dose of study drug during the treatment period.
Measure: Mean (Standard Deviation); unit: units on scale
Arm/Group | Dexlansoprazole 60 mg QD | Dexlansoprazole 60 mg BID
Number analyzed (Participants) | 3 | 3
units on scale
  Baseline | 7.3 (10.21) | 12.0 (10.00)
  Change at Month 12 | -3.0 (3.00) | -11.0 (8.54)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 30 days after last dose of study drug (Month 13).
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Dexlansoprazole 60 mg QD | Dexlansoprazole 60 mg BID
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/3
Other Adverse Events (participants affected / at risk) | 2/3 | 2/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexlansoprazole 60 mg QD (N=3) | Dexlansoprazole 60 mg BID (N=3)
Hypotension (Vascular disorders) | 0 | 1
Aspiration pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — The adverse event occurred postcolonoscopy.
Worsening of back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexlansoprazole 60 mg QD (N=3) | Dexlansoprazole 60 mg BID (N=3)
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.